CLINICAL TRIAL: NCT06077864
Title: A Phase 3, Randomised, Double-blind, Parallel-group, Event-driven, Cardiovascular Safety Study With BI 456906 Administered Subcutaneously Compared With Placebo in Participants With Overweight or Obesity With Established Cardiovascular Disease (CVD) or Chronic Kidney Disease, and/or at Least Two Weight-related Complications or Risk Factors for CVD
Brief Title: A Study to Test the Effect of Survodutide (BI 456906) on Cardiovascular Safety in People With Overweight or Obesity (SYNCHRONIZE™ - CVOT)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0040; 2022-502442-27-00 (Registry Identifier: CTIS); U1111-1289-0174 (Registry Identifier: WHO registry)
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- survodutide 3.6 mg (Experimental)
  Interventions: Drug: survodutide
- survodutide 6.0 mg (Experimental)
  Interventions: Drug: survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: survodutide — once weekly subcutaneous injection
  Other Names: BI 456906
  Arms: survodutide 3.6 mg; survodutide 6.0 mg
Drug: Placebo — once weekly subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 18 years old and have a body mass index (BMI) of 27 kg/m2 or more. People can take part if they have cardiovascular or chronic kidney disease. People who have at least 2 health problems related to their weight or risks of cardiovascular disease can participate. Participants must have previously tried to lose weight by changing their diet.

The purpose of this study is to find out whether people with overweight or obesity who take a medicine called survodutide (BI 456906) are less or more likely to develop serious cardiovascular problems. It also aims to find out whether health parameters like blood pressure improve. Overweight and obesity are linked to cardiovascular disease. Survodutide is a medicine that is developed to help people with obesity or overweight to lose weight.

Participants are divided into 3 groups of almost equal size. 2 groups get different doses of survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Every participant has a 2 in 3 chance of getting survodutide. Participants inject survodutide or placebo under the skin once a week. All participants also receive counselling on diet and physical activity.

Participants are in the study for up to 2 years and 3 months. During this time, it is planned that participants visit the study site up to 21 times and attend remote visits by video calls. During these visits, the doctors check participants' cardiovascular and overall health. The results are compared between survodutide and placebo groups. The study staff also takes note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years at the time of signing informed consent, and at least the legal age of consent in countries where it is >18 years.
2. Body mass index (BMI) ≥27 kg/m2 at screening with established cardiovascular disease (CVD) and/or at least 2 weight-related complications or risk factors for CVD OR BMI ≥30 kg/m2 at screening with established CVD or chronic kidney disease (CKD), and/or at least 2 weight-related complications or risk factors for CVD.

Further inclusion criteria apply.

Exclusion criteria:

1. Previous treatment with glucagon-like peptide-1 receptor (GLP-1R) agonists within 3 months before screening.
2. Type 1 diabetes.
3. Less than 3 months between the last dose of GLP-1R agonists and GLP-1R agonist/insulin/glucose-dependent insulinotropic polypeptide (GIP) combinations and screening.
4. Known clinically significant gastric emptying abnormality (e.g., severe diabetic gastroparesis or gastric outlet obstruction).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5531 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, non-fatal MI, ischaemia related coronary revascularisation, or HFE (to demonstrate non-inferiority) | up to Week 114
  Heart failure events (HFE) includes hospitalisation for heart failure (HHF), emergency room visit, urgent care visit, or urgent outpatient heart failure (HF) visit (5-point major adverse cardiac event (5P-MACE)) CV-Cardiovascular MI-Myocardial infarction

SECONDARY OUTCOMES:
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, or non-fatal MI (3-point major adverse cardiac event (3P-MACE)) (to demonstrate non-inferiority) | up to Week 114
Absolute change in systolic blood pressure (SBP) (mmHg) from baseline to Week 72 | Baseline and at Week 72
Absolute change in waist circumference (cm) from baseline to Week 72 | Baseline and at Week 72
Absolute change in Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) from baseline to Week 72 in trial participants with HF at baseline | At Baseline and at Week 72
  KCCQ-TSCC scale score range is from 0 to 100 where low score means patient not doing well and higher score means patient doing better.
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, non-fatal MI, ischaemia related coronary revascularisation, or HFE (to demonstrate superiority) | up to Week 114
Percentage change in body weight from baseline to Week 72 | Baseline and at Week 72
Absolute change in diastolic blood pressure (DBP) (mmHg) from baseline to Week 72 | Baseline and at Week 72
Absolute change in aspartate aminotransferase (AST) (U/L) from baseline to Week 72 | Baseline and at Week 72
Absolute change in alanine aminotransferase (ALT) (U/L) from baseline to Week 72 | Baseline and at Week 72
Absolute change in glycosylated haemoglobin A1c (HbA1c) (mmol/mol) from baseline to Week 72 in trial participants with type 2 diabetes mellitus (T2DM) | Baseline and at Week 72
Absolute change in HbA1c (%) from baseline to Week 72 in trial participants with T2DM | Baseline and at Week 72
Time to onset of T2DM in trial participants without T2DM at baseline | up to Week 114
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, non-fatal MI, or ischaemia related coronary revascularisation (4-point major adverse cardiac event (4P-MACE)) | up to Week 114
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, non-fatal MI, or HFE (3P-MACE+ HFE) | up to Week 114
Time to first occurrence of any of the adjudicated components of the composite endpoint consisting of: CV death, non-fatal stroke, or non-fatal MI (3P-MACE) | up to Week 114
Time to first occurrence of adjudicated CV death or adjudicated HFE | up to Week 114
Time to first occurrence of adjudicated CV death or adjudicated HHF | up to Week 114
Time to first occurrence of adjudicated HFE | up to Week 114
Time to adjudicated CV death | up to Week 114
Time to all-cause mortality | up to Week 114
Time to first occurrence of adjudicated non-fatal MI | up to Week 114
Time to first occurrence of adjudicated non-fatal stroke | up to Week 114
Time to first occurrence of adjudicated ischaemia related coronary revascularisation | up to Week 114
Achievement of body weight reduction ≥5% from baseline to Week 72 | Baseline and at Week 72
Achievement of body weight reduction ≥10% from baseline to Week 72 | Baseline and at Week 72
Achievement of body weight reduction ≥15% from baseline to Week 72 | Baseline and at Week 72
A composite of death, number of adjudicated HFEs, time to first adjudicated HFE and change from baseline in KCCQ-TSS at 72 weeks assessed by the win ratio in trial participants with HF at baseline | At baseline and at 72 Weeks
  Win ratio will be assessed as below:
  The primary efficacy endpoint will be analyzed using the clinical benefit approach comparing every participant in the BI 456906 arm to every participant in the placebo arm to determine a winner.
  A winner in the pair-wise comparison has a delayed time to the occurrence of death; if that cannot be determined, a winner has fewer HFEs; if the number of HFEs is the same a winner has a delayed time to the occurrence of first HFE; if that rule does not determine a winner, a winner has a more favorable (less increase or more decrease) change in KCCQ-CSS between baseline and at 72 weeks, otherwise the pair will be recorded as tied. The estimated net benefit (win ratio is then calculated as the total number of wins in the BI 456906 group across all strata divided by the total number of losses) will be provided.
  KCCQ-TSCC scale score range is from 0 to 100 where low score means patient not doing well and higher score means patient doing better.

CONTACTS AND LOCATIONS:
Locations (539):
- United States (153):
  - Cardiology P.C., Birmingham, Alabama
  - AMR Daphne, Daphne, Alabama
  - AMR Mobile, Mobile, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - The Institute for Liver Health II DBA Arizona Clinical Trials, Chandler, Arizona
  - Clinical Research Institute of Arizona, LLC, Sun City West, Arizona
  - AMR Phoenix, Tempe, Arizona
  - Arizona Liver Health-Tucson-67516, Tucson, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Velocity Clinical Research-Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Velocity Clinical Research - Los Angeles, Los Angeles, California
  - Catalina Research Institute, LLC - Montclair, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - NorthBay Clinical Research, LLC, Santa Rosa, California
  - Velocity Clinical Research-Van Nuys-70286, Van Nuys, California
  - Peak Gastroenterology Associates-Colorado Springs-62256, Colorado Springs, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Proactive Clinical Research, Boca Raton, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Nature Coast Clinical Research-Crystal River-62355, Crystal River, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - AMR Fort Myers, Fort Myers, Florida
  - Covenant Metabolic Specialists, LLC - Fort Myers, Fort Myers, Florida
  - Velocity Clinical Research-Hallandale Beach-67888, Hallandale, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Clinical Site Partners LLC, Leesburg, Florida
  - Suncoast Research Group, Miami, Florida
  - Verus Clinical Research Corporation, Miami, Florida
  - Clinical Trial Services, Corp, Miami, Florida
  - Synexus-Pinellas Park-69294, Pinellas Park, Florida
  - East Coast Institute for Research, LLC-Saint Augustine-63032, Saint Augustine, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Santos Research Center, Corp., Tampa, Florida
  - Covenant Metabolic Specialists, LLC - Sarasota, University Park, Florida
  - Javara-Albany-67356, Albany, Georgia
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - Javara-Fayetteville-67354, Fayetteville, Georgia
  - NSC Research Inc, Johns Creek, Georgia
  - The Jones Center Clinical Research, LLC, Macon, Georgia
  - Urban Family Practice Associates, PC, Marietta, Georgia
  - Javara-Savannah-67450, Savannah, Georgia
  - Endeavor Health Clinical Operations - Northwest Community Healthcare, Arlington Heights, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - Research by Design, LLC, Chicago, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - AMR El Dorado, El Dorado, Kansas
  - AMR Newton, Newton, Kansas
  - AMR Wichita East, Wichita, Kansas
  - Research Integrity, LLC, Owensboro, Kentucky
  - Grace Research, LLC-Bossier City-51040, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - AMR New Orleans, New Orleans, Louisiana
  - Grace Research, LLC-Shreveport-64616, Shreveport, Louisiana
  - Javara Inc.-Annapolis-68997, Annapolis, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Domino's Farms, Ann Arbor, Michigan
  - Elite Research Center, LLC, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The National Diabetes & Obesity Research Institute, Diamondhead, Mississippi
  - Prime Health and Wellness, Fayette, Mississippi
  - Velocity Clinical Research-Gulfport-68930, Gulfport, Mississippi
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Skyline Medical Center, Elkhorn, Nebraska
  - Methodist Physicians Clinic, Fremont, Nebraska
  - AMR Las Vegas, Las Vegas, Nevada
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - NJ Heart LLC, Linden, New Jersey
  - IMA Clinical Research-Warren-69742, Warren Township, New Jersey
  - IMA Clinical Research Albuquerque, Albuquerque, New Mexico
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - Synexus Clinical Research US, Inc., New York, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Accellacare of Cary, Cary, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Javara-Charlotte-67884, Charlotte, North Carolina
  - Accellacare-Mooresville-69123, Mooresville, North Carolina
  - Lucas Research, New Bern, North Carolina
  - Wake Forest University Health Sciences-Winston-Salem-69719, Winston-Salem, North Carolina
  - Velocity Clinical Research-Cincinnati-69044, Cincinnati, Ohio
  - Synexus Clinical Research-Columbus-69427, Columbus, Ohio
  - Centricity Research-Columbus-68879, Columbus, Ohio
  - Aventiv Research Inc.-Dublin-62009, Dublin, Ohio
  - Clinical Research Institute of Ohio, LLC, Westlake, Ohio
  - Tekton Research-Edmond-68875, Edmond, Oklahoma
  - AMR Norman, Norman, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Velocity Clinical Research-Medford-69053, Medford, Oregon
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Tristar Clinical Investigations PC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians-Pittsburgh-63932, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians-Uniontown-69137, Uniontown, Pennsylvania
  - Velocity Clinical Research-East Greenwich-68873, East Greenwich, Rhode Island
  - Synexus - Anderson, Anderson, South Carolina
  - Velocity Clinical Research-Anderson-69093, Anderson, South Carolina
  - Velocity Clinical Research-Gaffney-69046, Gaffney, South Carolina
  - Tribe Clinical Research LLC, Greenville, South Carolina
  - Velocity Clinical Research-Greenville-69045, Greenville, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Velocity Clinical Research-Union-68888, Union, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Alliance for Multispecialty Research, LLC-Knoxville-69693, Knoxville, Tennessee
  - Accellacare of Knoxville-Knoxville-69135, Knoxville, Tennessee
  - Accellacare of Knoxville-Knoxville-69714, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc-Memphis-65988, Memphis, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Headlands Research, Brownsville, Texas
  - Privia Medical Group Gulf Coast, PLLC, Conroe, Texas
  - Velocity Clinical Research-Dallas-69170, Dallas, Texas
  - Javara Inc. - Fort Worth, Fort Worth, Texas
  - Houston Research Institute, Houston, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Tekton Research-San Antonio-68916, San Antonio, Texas
  - Javara Inc. and Privia Medical Group Gulf Coast, PLLC, San Marcos, Texas
  - Javara Inc.-Stephenville-68996, Stephenville, Texas
  - DM Clinical Research - Martin Diagnostic Clinic, Tomball, Texas
  - Velocity Clinical Research, Waco, Waco, Texas
  - Physicians' Research Options. LLC, Draper, Utah
  - Alliance for Multispecialty Research, LLC-Layton-69691, Layton, Utah
  - Synexus Clinical Research-Salt Lake City-69293, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Velocity Clinical Research-West Jordan-69043, West Jordan, Utah
  - Washington Center for Weight Management and Research, Inc., Arlington, Virginia
  - Seven Corners Medical Center, Falls Church, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Selma Medical Associates, Winchester, Winchester, Virginia
  - Velocity Clinical Research-Seattle-69881, Seattle, Washington
  - Velocity Clinical Research-Spokane-69716, Spokane, Washington
  - Clinical Investigation Specialists, Inc.-Kenosha-69111, Kenosha, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Argentina (14):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Mautalen- Salud e Investigacion, CABA
  - Centro Medico Dra Laura Maffei, Ciudad Autonoma Buenos Aires
  - Glenny Corp. S.A. Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Centro Medico Viamonte, Ciudad Autonoma de Bs As
  - Sanatorio Güemes, Ciudad Autonoma de Bs As
  - Consultorio de Investigacion Clinica EMO SRL, Ciudad Autonoma de Buenos Aire
  - CIPREC, Ciudad Autonoma de Buenos Aire
  - CIDIM - Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Hospital Privado - Centro Medico de Cordoba S.A., Parque Velez Sarsfield
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (11):
  - The Boden Initiative, Camperdown, New South Wales
  - Novatrials, Charlestown, New South Wales
  - Royal North Shore Hospital-St Leonards-66471, St Leonards, New South Wales
  - Momentum Clinical Research - Taringa, Taringa, Queensland
  - Momentum Clinical Research Taringa, Wellers Hill, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Advara Heart Care-Leabrook-69072, Leabrook, South Australia
  - Victorian Heart Hospital, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Advara Heart Care-Joondalup-69073, Joondalup, Western Australia
  - Southern Adelaide Diabetes & Endocrine services, Oaklands Park
- Austria (8):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Convent Hospital Barmherzige Brüder, Linz
  - LKH Salzburg University Hospital, Salzburg
  - Hospital Stockerau, Stockerau
  - Klinik Landstrasse, Vienna
  - Private Practice - Dr. Ursula Hanusch-Enserer, Vienna
  - AKH - Medical University of Vienna, Vienna
- Belgium (3):
  - AZ Sint-Jan Brugge, Bruges
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
- Brazil (12):
  - Hospital Universitário João de Barros Barreto, Belém
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília
  - Chronos Pesquisa Clinica, Brasília
  - Cline Research Center, Curitiba
  - Instituto de Estudos e Pesquisas Clínicas IEP-CE, Fortaleza
  - Instituto Brasil de Pesquisa Clinica (IBPClin), Rio de Janeiro
  - ISPEM - Instituto São Jose dos Campos em Pesquisas Medicas, São José dos Campos
  - Irmandade da Santa Casa de Misericórdia de São Paulo - IPEC - Instituto de Pesquisa Clínica, São Paulo
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - BR Trials, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo
- Bulgaria (14):
  - MHAT "Yuliya Vrevska" EOOD, Byala, Byala
  - MHAT - Dobrich, AD, Dobrich
  - Multy profile hospital for active treatment Sv.Ivan Rilski, Dupnitsa
  - Multiprofile Hospital for Active Treatment Trimontsium OOD, Plovdiv
  - MHAT "St. Caridad", Plovdiv
  - Multy Profile Hospital for active treatment Hadzhi Dimirar, Sliven
  - Diagnostic & Consultancy Center "Ascendent", Sofia, Sofia
  - Alexandrovska University Hospital, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - ASOMHIDC - Individual practice "Cardio Tonus" EOOD, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
  - Medical Center Berbatov, Yambol
  - MHAT St Panteleimon, Yambol
- Canada (25):
  - Richmond Road Diagnostic & Treatment Centre, Calgary, Alberta
  - C-ENDO Diabetes & Endocrinology Clinic, Calgary, Alberta
  - CARe Clinic (Red Deer), Red Deer, Alberta
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Centricity Research (Brampton), Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Centricity Research (Etobicoke), Etobicoke, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc., Hamilton, Ontario
  - Western Centre for Public Health & Family Medicine (LHRI), London, Ontario
  - Centricity Research (Oshawa), Oshawa, Ontario
  - Bluewater Clinical Research, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Centricity Research (Bayview), Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Clinical Research Solutions Inc. (Waterloo), Waterloo, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Centre de Medecine Metabolique de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
  - Recherche Clinique Sigma Inc., Québec
- China (34):
  - Beijing Chao-Yang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - Changzhou Second People's Hospital, Changzhou
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Hangzhou First People's Hospital, Hangzhou
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of University of South China, Hengyang
  - Huai'an first people's hospital, Huai'an
  - Huzhou Central Hospital, Huzhou
  - Center Hospital of Jinan, Jinan
  - Lishui Municipal Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Nanchang People's Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - First Hospital of Qinhuangdao, Qinhuangdao
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Shanghai Pudong New District People's Hospital, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Suzhou Science & Technology Town Hospital, Suzhou
  - Shaanxi Provincial People's Hospital, Xi'an
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - Xianyang Hospital of Yan'an University, Xianyang
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Czechia (12):
  - St. Anna Hospital, Brno
  - DIKa centrum s.r.o., Havířov
  - Center for Osteoporosis Therapy, Karlovy Vary
  - Internal and Diabetes Clinic, Náchod
  - PreventaMed, s.r.o., Olomouc
  - University Hospital Ostrava, Ostrava-Poruba
  - Internal ambulance Dialine s.r.o., Pilsen
  - Synexus Czech s.r.o., Prague
  - General Faculty Hospital, Prague, Prague
  - OB Klinika, Prague
  - Institute for Clinical and Experimental Medicine-Prague-66083, Prague
  - ResTrial s.r.o., Prague
- Denmark (5):
  - Aarhus University Hospital, Aarhus N
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Hvidovre Hospital, Hvidovre
- Finland (5):
  - CRST Helsinki Oy, Helsinki
  - StudyCor Oy, Jyväskylä
  - Terveystalo Pori Lääkäritalo, Pori
  - Tampere University Hospital, Tampere
  - Terveystalo Pulssi, Turku, Turku
- Germany (20):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Velocity Clinical Research Germany GmbH, Berlin, Berlin
  - DRK Kliniken Berlin Köpenick, Berlin
  - Synexus Clinical Research GmbH, Berlin, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Synexus Clinical Research GmbH, Frankfurt, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - St. Josefskrankenhaus Heidelberg, Heidelberg
  - Universität des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Synexus Clinical Research GmbH, Leipzig, Leipzig
  - Velocity Clinical Research Germany GmbH, Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Westfälische Wilhelms-Universität Münster, Münster
  - CEDA Research GBR, Pohlheim
  - Universitätsklinikum Tübingen, Tübingen
- Greece (9):
  - General Hospital of Athens "Laiko", Athens
  - Attikon University Hospital, Haidari-Athens
  - University General Hospital of Heraklion, Heraklion, Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - Iatriko of Athens Group/ Iatriko of P. Faliro, P. Faliro
  - Iatriko Psychikou, Psychikó
  - Gen. Hosp. of Thessaloniki "Hippokation", Department of Endocrinology, Thessaloniki
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Hong Kong (3):
  - Prince of Wales Hospital-Hong Kong-20715, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong
- Hungary (15):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Obudai Egeszegugyi Centrum Kft., Budapest
  - Synexus Hungary Healthcare Service Ltd., Budapest
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Bajcsy-Zsilinszky Hospital and Clinic, Budapest
  - Semmelweis University, Budapest
  - University Debrecen Hospital, Debrecen
  - Erzsebet Nursing Home, Gödöllő
  - Synexus Hungary Healthcare Service Ltd, Gyula
  - Trial Pharma Kft, Gyula
  - BKS Research Ltd, Hatvan
  - Studium Egeszseghaz Kft., Kalocsa
  - Somogy County Kaposi Mor Teaching Hospital, Kaposvár
  - Obudai Egeszegugyi Centrum, Zalaegerszeg
  - SYNEXUS Hungary Health Care Services Ltd-Zalaegerszeg-69406, Zalaegerszeg
- India (8):
  - Kamalnayan Bajaj Hospital, Aurangabad
  - S.P. Medical College & Associated Group of Hospitals, Bikaner
  - Apollo Speciality Hospital, Chennai
  - LPS Institute of Cardiology, Kanpur
  - Shrikrishna Hrudayalaya and Critical Care Centre, Maharashtra
  - Batra Hospital and Medical Research Centre, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Shri B.D. Mehta Mahavir Heart Institute, Surat
- Ireland (2):
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
- Italy (10):
  - Humanitas Gavazzeni, Bergamo
  - Ospedale S.M. Goretti, Latina
  - IRCCS MultiMedica, Milan
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Policlinico "Paolo Giaccone", Palermo
  - Università Campus Bio-Medico - ROMA, Roma
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - A.O.U. Senese, Siena
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Torino
- Japan (24):
  - Meitetsu Hospital, Aichi, Nagoya
  - Nagoya Kyoritsu Hospital, Aichi, Nagoya
  - Chubu Rosai Hospital, Aichi, Nagoya
  - Daido Clinic, Aichi, Nagoya
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Takagi Hospital, Fukuoka, Okawa
  - Seino Internal Medicine Clinic, Fukushima, Koriyama
  - Iryouhouijneiwakai Minamiakatsuka Clinic, Ibaraki, Mito
  - Matsuba Clinic, Kanagawa, Kawasaki
  - Sagamihara Kyodo Hospital, Kanagawa, Sagamihara
  - Saiseikai Yokohamashi Nanbu Hospital, Kanagawa, Yokohama
  - Takeshita Hospital, Kochi, Kochi
  - Kyoto Okamoto Memorial Hospital, Kyoto, Kuse-gun
  - Sato Hospital, Miyagi, Sendai
  - Urasoe General Hospital, Okinawa, Urasoe
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - Saiseikai Kawaguchi Hospital, Saitama, Kawaguchi
  - Koshigaya Municipal Hospital, Saitama, Koshigaya
  - Saitama Sekishikai Hospital, Saitama, Sayama
  - Sayama General Clinic, Saitama, Sayama
  - Omihachiman Community Medical Center, Shiga, Omihachiman
  - Minamino Cardiovascular Hospital, Tokyo, Hachioji
  - NewHeart Watanabe Institute, Tokyo, Suginami-ku
  - Saiseikai Wakayama Hospital, Wakayama, Wakayama
- Kazakhstan (4):
  - Institute of Gastroenterology, Gepatology and Metabolism LLP, Almaty
  - Academy of Preventive Medicine, Clinic "Vitalem", Almaty
  - Multidisciplinary City Hospital №1 of the Akimat of Astana, Astana
  - National Research Medical Center (NNMC), Astana
- Mexico (6):
  - Medical Center Metas S.C., Chihuahua City
  - Instituto de Diabetes, Obesidad y Nutrición S.C., Cuernavaca
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Clinica Omega Diabetes, Mexico City
  - CEDOPEC-Ctro Esp en Diab, Obesidad y Prev de Enf Cardiovasc, México
  - Cardiolink Clin Trials S.C., Monterrey
- Netherlands (4):
  - Rijnstate Hospital, Arnhem
  - Spaarne Ziekenhuis, Haarlem
  - Diakonessenhuis Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
- New Zealand (7):
  - P3 Research Palmerston North, Palmerston North, Migration Data
  - Optimal Clinical Trials, Auckland
  - Pacific Clinical Research Network - Forte Christchurch, Christchurch
  - Momentum Clinical Research, Lower Hutt
  - Middlemore Clinical Trials, Papatoetoe
  - Pacific Clinical Research Network - Rotorua, Rotorua
  - P3 Research Kapiti, Waikanae Beach
- Norway (4):
  - Vestre Viken HF, Drammen Sykehus, Drammen
  - Akershus Universitetssykehus HF, Lørenskog
  - St. Olavs Hospital, Universitetssykehuset i Trondheim, Trondheim
  - Sykehuset i Vestfold, Avd. Tønsberg, Tønsberg
- Poland (34):
  - Medical University of Bialystok, Bialystok
  - Trial Medica, Bialystok
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - NZOZ Medical Center KERmed, Bydgoszcz
  - Synexus Poland, Branch in Czestochowa, Częstochowa
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Gdynia
  - Przychodnie Grudziadz sp.zo.o, Grudziądz
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Katowice
  - Silmedic Sp. z o.o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Salvia Lekston I Madej Sp. J., Katowice
  - Diab-Endo-Met Medical Center, Krakow
  - Unicardia Specialist Medical Center, Krakow
  - Synexus Lodz Medical Center, Lodz
  - Med-Gastr Medical Center, Lodz
  - Clinical Best Solutions, Lublin
  - Ekamed Sp. z o.o., Lublin
  - Futuremeds Sp. z o.o. Olsztyn, Olsztyn
  - Synexus Poland, Branch in Poznan, Poznan
  - Metabolic Health Center Pawel Bogdanski, Poznan
  - Private Practice Dr. Ewa Krzyzagorska, Poznan
  - Padre Pio Regional Hospital in Przemysl, Przemyśl
  - Centrum Medyczne Medyk, Rzeszów
  - Velocity Skierniewice Sp. z o.o., Skierniewice
  - NZOZ Procordis, Cardiology Research Center of Sopot, Sopot
  - Velocity Staszow, Staszów
  - DC-MED, Swidnica
  - Clinical Best Solutions Sp. z o.o. S.K., Warsaw
  - NBR Polska, Warsaw
  - National Medical Institute MSWiA, Warsaw
  - Centrum Medyczne Synexus, Warsaw
  - ETG Warszawa, Warsaw
  - Synexus Poland, Branch in Wroclaw, Wroclaw
- Portugal (12):
  - Hospital de Cascais Dr. José de Almeida, Alcabideche
  - ULS da Região de Aveiro, Aveiro
  - ULS Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS do Alto Ave, Guimarães
  - ULS de São José, Lisbon
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Hospital da Luz, Lisbon
  - Cardiolima - Centro Diagnostico Cardio-pulmonar de Ponte de Lima, Lda., Ponte de Lima
  - ULS de Entre Douro e Vouga, Santa Maria da Feira
  - UCARDIO, Torres Novas
  - Hospital da Luz Arrábida, Vila Nova de Gaia
- Puerto Rico (2):
  - Advanced Clinical Research, Bayamón
  - Ponce School of Medicine/CAIMED Center, Ponce
- Saudi Arabia (4):
  - King Fahad Specialist Hospital - Research Center, Dammam
  - King AbdulAziz University Hospital, Jeddah
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Saud Medical City, Riyadh
- Slovakia (6):
  - METABOL KLINIK s.r.o., Bratislava, Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava, Bratislava
  - Medical Group Kosice s.r.o, Košice
  - IN-DIA s.r.o., Lucenec, Lučenec
  - Funkystuff s.r.o., Nové Zámky
  - DIAB sro, Rožňava
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (15):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Dr. Peset, Valencia
- Taiwan (5):
  - Chang-Hua Christian Hospital, Changhua
  - Chia-Yi Christian Hospital, Chia-Yi City
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (13):
  - Adana City Hospital, Adana
  - Baskent University Hospital, Adana
  - Akdeniz UTF Endokrinoloji ve Metabolizma Hastaliklari BD, Antalya
  - Inonu Uni. Med. Fac., Battalgazi, Battalgazi
  - Bursa Yuksek Ihtisas EAH, Bursa
  - Dicle Universitesi Tip Fakultesi, Diyarbakır
  - Koc Universitesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi-Istanbul-1433, Istanbul
  - Acibadem Universitesi Atakent Hastanesi, Istanbul
  - İstanbul Prof.Dr. Cemil Taşçıoğlu City Hospital, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Marmara Universitesi Tip Fakultesi, Istanbul
  - Zonguldak Bulent Ecevit UTF, Zonguldak
- United Kingdom (22):
  - University Hospital Monklands, Airdrie
  - Antrim Area Hospital, Antrim
  - Waterloo Medical Centre, Blackpool
  - Synexus - Cardiff, Cardiff
  - Synexus - Lancashire, Chorley
  - Ninewells Hospital & Medical School, Dundee
  - Synexus - Midlands, Edgbaston
  - Wellcome Trust Clinical Research Facility, Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Synexus - Glasgow, Glasgow
  - Synexus - Hexham, Hexham
  - Leicester General Hospital, Leicester
  - Lincoln County Hospital, Lincoln
  - Synexus - Merseyside, Liverpool
  - William Harvey Research Limited, London
  - Altnagelvin Area Hospital, Londonderry
  - Manchester Royal Infirmary, Manchester
  - Synexus - Manchester, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - FutureMeds - Newcastle, Newcastle upon Tyne
  - Swansea University Medical School, Swansea
  - University Hospital Wishaw, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- [Derived] Kosiborod MN, Platz E, Wharton S, le Roux CW, Brueckmann M, Ajaz Hussain S, Unseld A, Startseva E, Kaplan LM; SYNCHRONIZE-CVOT Trial Committees and Investigators. Survodutide for the Treatment of Obesity: Rationale and Design of the SYNCHRONIZE Cardiovascular Outcomes Trial. JACC Heart Fail. 2024 Dec;12(12):2101-2109. doi: 10.1016/j.jchf.2024.09.004. Epub 2024 Oct 23. PMID 39453356
- See also: Related Info — http://www.mystudywindow.com